CLINICAL TRIAL: NCT00519961
Title: A Prospective Study to Assess the Screening Value of N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP) for the Identification of Patients That Benefit From Additional Cardiac Testing Prior to Vascular Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD000485; DECREASE-VI
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

ARMS (2):
- A (Experimental)
  Interventions: Device: Elecsys®proBNP
- B (Experimental)
  Interventions: Device: Elecsys®proBNP

INTERVENTIONS:
Device: Elecsys®proBNP

SUMMARY:
The purpose of this study is to validate the screening potential of NT-proBNP for the identification of patients scheduled for vascular surgery who would benefit from additional pre-operative cardiac testing. All patients will have NT-proBNP concentrations measured pre-operatively. For low-intermediate risk patients only those with abnormal values will receive further cardiac testing; all high risk patients will be referred for additional testing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥18 years of age
* Patients with peripheral vascular atherosclerosis, scheduled for vascular surgery

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2007-02; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Collection of 30-day and 1-year postoperative cardiac events | 30-day and 1-year postoperation

CONTACTS AND LOCATIONS:
Overall Officials: Wilma Verhagen-Kamerbeek, Study Director — Roche Diagnostics GmbH
Locations (2):
- Dublin, Ireland
- Rotterdam, Netherlands